CLINICAL TRIAL: NCT07312370
Title: Intravenous Esomeprazole Combined With Sucralfate Suspension for Ulcer Healing and Complication Prevention After Gastric Endoscopic Submucosal Dissection: A Prospective, Randomized, Controlled Trial
Brief Title: Esomeprazole Plus Sucralfate for Post-ESD Ulcer Healing: A Randomized Controlled Trial
Acronym: ESUS-ESD
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: LanZhou University (Other)
Responsible Party: Principal Investigator, Zhaofeng Chen, Clinical Professor, LanZhou University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LDYYczf2025121701
Record Dates: First submitted 2025-12-17; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Early Gastric Cancer; Gastric Dysplasia; Gastric Neoplasms; Peptic Ulcer With Haemorrhage; Gastric Ulcer
Keywords: Endoscopic Submucosal Dissection; Gastric Cancer; Ulcer Healing; Proton Pump Inhibitor; Post-ESD Ulcer; Early Gastric Neoplasm
MeSH Terms: conditions — Stomach Neoplasms; Peptic Ulcer Hemorrhage; Stomach Ulcer | interventions — Esomeprazole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: This is an open-label study for participants and care providers due to the nature of oral suspension that cannot be easily matched with placebo. However, outcome assessors (endoscopists evaluating images and videos) and data analysts will be blinded to treatment allocation until database lock.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Esomeprazole + Sucralfate (Intervention Group) (Experimental): * Days 1-3: Esomeprazole 40mg intravenously every 12 hours
  * Days 4-56: Esomeprazole 40mg orally once daily (before breakfast) + Sucralfate suspension 1g orally twice daily (1 hour before breakfast and at bedtime on empty stomach)
  Interventions: Drug: Esomeprazole (Intravenous); Drug: Esomeprazole (Oral); Drug: Sucralfate Suspension; Procedure: Gastric Endoscopic Submucosal Dissection (ESD)
- Esomeprazole Alone (Control Group) (Active Comparator): * Days 1-3: Esomeprazole 40mg intravenously every 12 hours
  * Days 4-56: Esomeprazole 40mg orally once daily (before breakfast)
  Interventions: Drug: Esomeprazole (Intravenous); Drug: Esomeprazole (Oral); Procedure: Gastric Endoscopic Submucosal Dissection (ESD)

INTERVENTIONS:
Drug: Esomeprazole (Intravenous) — Esomeprazole 40mg intravenously every 12 hours for 3 days (Days 1-3 post-ESD)
  Other Names: Esomeprazole Sodium
Drug: Esomeprazole (Oral) — Esomeprazole 40mg orally once daily, taken before breakfast, for 8 weeks (Days 4-56)
  Other Names: Esomeprazole Magnesium
Drug: Sucralfate Suspension — Sucralfate suspension 1g (one sachet) orally twice daily for 8 weeks. Administered 1 hour before breakfast and at bedtime on empty stomach (2-3 hours after dinner). Should be taken separately from other medications (≥1-2 hours apart).
  Arms: Esomeprazole + Sucralfate (Intervention Group)
Procedure: Gastric Endoscopic Submucosal Dissection (ESD) — Standardized gastric ESD procedure including lesion marking, submucosal injection, circumferential incision, submucosal dissection, and complete coagulation of all visible vessels at the ulcer base.

SUMMARY:
Endoscopic submucosal dissection (ESD) is an established treatment for early gastric cancer and precancerous lesions. Post-ESD artificial ulcers may lead to complications including delayed bleeding (3-15%) and prolonged healing. Current guidelines recommend high-dose proton pump inhibitors (PPIs), but evidence for additional mucosal protective agents remains limited.

This study aims to evaluate whether combining sucralfate suspension with standard intravenous esomeprazole therapy improves ulcer healing and reduces complications after gastric ESD compared to esomeprazole alone.

This is a prospective, randomized, controlled, outcome-assessor-blinded trial. A total of 120 patients undergoing gastric ESD will be randomly assigned 1:1 to receive either:

* Intervention group: Intravenous esomeprazole 40mg twice daily (3 days) followed by oral esomeprazole 40mg once daily PLUS sucralfate suspension 1g twice daily for 8 weeks
* Control group: Intravenous esomeprazole 40mg twice daily (3 days) followed by oral esomeprazole 40mg once daily for 8 weeks The primary outcome is ulcer reduction rate at 4 weeks post-ESD, assessed by endoscopy. Secondary outcomes include complete ulcer healing rate at 8 weeks, delayed bleeding rate, symptom scores, and safety parameters.

This study will provide high-quality evidence regarding the role of sucralfate as an adjunctive therapy for post-ESD ulcer management and may inform future clinical guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years, male or female
2. Diagnosed with early gastric cancer or high-grade intraepithelial neoplasia planned for gastric ESD
3. Lesion location: Gastric corpus, antrum, or angle (cardiac lesions may be included but will require subgroup analysis)
4. Successful en bloc resection achieved by ESD
5. Post-ESD artificial ulcer diameter ≥2 cm
6. Complete coagulation of all visible vessels during ESD procedure
7. ECOG performance status 0-1
8. Able to comply with follow-up visits and endoscopic examinations
9. Voluntary participation with written informed consent

Exclusion Criteria:

1. Previous gastric surgery history
2. Active peptic ulcer disease (confirmed by pre-ESD endoscopy) within 1 month
3. Recent upper gastrointestinal bleeding (within 1 month, excluding tumor-related bleeding)
4. Severe heart, liver, or kidney dysfunction (Child-Pugh class C, NYHA class III-IV, or CKD stage 4-5)
5. Coagulation disorders (INR >1.5 or platelet count <50×10⁹/L)
6. Uncontrolled diabetes (HbA1c >9%)
7. Known allergy or hypersensitivity to PPIs or sucralfate
8. Use of PPIs, H2 receptor antagonists, or mucosal protective agents within 2 weeks prior to ESD
9. Long-term anticoagulant therapy that cannot be discontinued (e.g., warfarin, direct oral anticoagulants)
10. Long-term NSAIDs or aspirin (>100mg/day) that cannot be discontinued
11. Unsuccessful complete (en bloc) resection (piecemeal resection)
12. Intraoperative perforation
13. Uncontrolled active bleeding during ESD
14. Pregnancy or lactation
15. Women of childbearing potential not using adequate contraception
16. Concurrent participation in another clinical trial
17. Any condition that, in the investigator's opinion, makes the patient unsuitable for study participation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2026-11-20 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Ulcer Reduction Rate at 4 Weeks Post-ESD | 4 weeks after ESD procedure (±3 days)
  The percentage reduction in ulcer area from baseline (immediately post-ESD) to 4 weeks, calculated as: Ulcer Reduction Rate (%) = [(Baseline ulcer area - Week 4 ulcer area) / Baseline ulcer area] × 100

SECONDARY OUTCOMES:
Ulcer Reduction Rate at 8 Weeks Post-ESD | 8 weeks after ESD procedure (±3 days)
  Same calculation method as primary outcome, assessed at 8 weeks
Ulcer Stage at 4 Weeks (Sakita Classification) | 4 weeks after ESD procedure (±3 days)
  Classification of ulcer healing stage according to Sakita classification: A1 (active with thick coat), A2 (healing with thinning coat), H1 (healing with regenerating epithelium, red), H2 (healing with thickened epithelium, red fading), S1 (scar stage, red), S2 (scar stage, white). Assessed by blinded endoscopists.
Complete Ulcer Healing Rate at 8 Weeks | 8 weeks after ESD procedure (±3 days)
  Proportion of patients achieving complete ulcer healing defined as scar stage (S1 or S2) on Sakita classification at 8 weeks post-ESD
Incidence of Delayed Bleeding | From 24 hours post-ESD up to 8 weeks
  Occurrence of delayed post-ESD bleeding defined as: hematemesis or melena accompanied by hemoglobin decrease ≥2 g/dL, or requiring blood transfusion or endoscopic hemostatic intervention. Time of bleeding occurrence will be recorded.
Change in Epigastric Pain Score | Baseline (Day 0), Day 7, Week 4, and Week 8
  Severity of epigastric pain assessed using Visual Analog Scale (VAS) ranging from 0 (no pain) to 10 (worst imaginable pain). Change from baseline at each time point will be calculated.
Change in Bloating Score | Baseline (Day 0), Day 7, Week 4, and Week 8
  Severity of bloating assessed using Visual Analog Scale (VAS) ranging from 0 (no bloating) to 10 (worst imaginable bloating). Change from baseline at each time point will be calculated.
Change in Acid Reflux Score | Baseline (Day 0), Day 7, Week 4, and Week 8
  Severity of acid reflux assessed using Visual Analog Scale (VAS) ranging from 0 (no reflux) to 10 (worst imaginable reflux). Change from baseline at each time point will be calculated.
Change in Quality of Life Score | Baseline (Day 0), Week 4, and Week 8
  Quality of life assessed using EQ-5D-5L questionnaire, which evaluates five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) with five levels each, plus a visual analog scale (0-100). Change from baseline will be calculated.
Rate of Rehospitalization Due to ESD-Related Complications | From Day 0 through Week 8
  Proportion of patients requiring rehospitalization due to post-ESD complications including delayed bleeding, severe pain, or other ESD-related adverse events
Need for Endoscopic Hemostatic Intervention | From Day 0 through Week 8
  Proportion of patients requiring emergency or urgent endoscopic hemostatic procedures (such as hemoclipping, coagulation, or injection therapy) for post-ESD bleeding
Incidence of Adverse Events | From Day 0 through Week 8
  Frequency and severity of all adverse events and serious adverse events, categorized by organ system and graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Medication Compliance Rate | Throughout 8-week treatment period
  Percentage of prescribed medication doses actually taken by the patient, calculated as: (Actual medication days / Expected medication days) × 100%. Assessed using medication diary and pill/sachet count. Compliance ≥80% will be considered good.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Lanzhou University, Lanzhou, Gansu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Takeuchi T, Ota K, Harada S, Edogawa S, Kojima Y, Tokioka S, Umegaki E, Higuchi K. The postoperative bleeding rate and its risk factors in patients on antithrombotic therapy who undergo gastric endoscopic submucosal dissection. BMC Gastroenterol. 2013 Sep 6;13:136. doi: 10.1186/1471-230X-13-136. PMID 24010587
- [Background] Tanaka S, Terasaki M, Kanao H, Oka S, Chayama K. Current status and future perspectives of endoscopic submucosal dissection for colorectal tumors. Dig Endosc. 2012 May;24 Suppl 1:73-9. doi: 10.1111/j.1443-1661.2012.01252.x. PMID 22533757
- [Background] Pimentel-Nunes P, Libanio D, Bastiaansen BAJ, Bhandari P, Bisschops R, Bourke MJ, Esposito G, Lemmers A, Maselli R, Messmann H, Pech O, Pioche M, Vieth M, Weusten BLAM, van Hooft JE, Deprez PH, Dinis-Ribeiro M. Endoscopic submucosal dissection for superficial gastrointestinal lesions: European Society of Gastrointestinal Endoscopy (ESGE) Guideline - Update 2022. Endoscopy. 2022 Jun;54(6):591-622. doi: 10.1055/a-1811-7025. Epub 2022 May 6. PMID 35523224